CLINICAL TRIAL: NCT06386796
Title: Renal Resistive Index as a Predictor of Acute Renal Impairment in High-risk Patients Admitted to Surgical Intensive Care Unit.
Brief Title: Renal Resistive Index as a Predictor of Acute Renal Impairment in High-risk Patients
Status: Recruiting | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Soudy Salah Hammad, Lecturer of anesthesia and surgical intensive care, Aswan University
Other Study IDs: Asw.U./867/11/23
Record Dates: First submitted 2024-04-04; First posted 2024-04-26 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Injury; Critical Illness
Keywords: renal resisitive index; surgical ICU; Cystatin C
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To study the ability of RRI, measured by bedside Doppler ultrasound, in detecting acute kidney injury in high-risk patients admitted to surgical intensive care unit, Aswan university hospital, compared with renal biomarkers and conventional assessment using urine output and serum creatinine levels.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common clinical problem encountered in critically ill patients, frequently in the setting of multiple organ failure, and is an independent risk factor for increase hospital stay and mortality risk.

Early-stage acute kidney injury was first assessed based on the risk, injury, failure, loss and end-stage (RIFLE) criteria in 2004, and then by the Acute Kidney Injury Network (AKIN) criteria in 2007. The Kidney Disease: Improving Global Outcomes (KDIGO) classification, based on both the AKIN and RIFLE criteria, was introduced in 2012, offering an assessment based on baseline creatinine and urine output.

The best strategy in clinical practice is to identify AKI as early as possible, reverse its cause, and even improve the sequelae. In the past decades, several serum creatinine (SCr)-based classification systems have been proposed to define AKI.

The limitations of SCr is that the determinants of SCr (rate of production, apparent volume of distribution, and rate of elimination) are variable. Therefore, there is an unmet need for other objective measures to help detect AKI in a timely manner. The role of several biomarkers in the early prediction or risk assessment of AKI has been proposed, including kidney tubular damage markers (e.g., neutrophil gelatinase-associated lipocalin (NGAL), kidney injury molecule-1 (KIM- 1), liver-type fatty acid-binding protein (L-FABP) and cystatin C).

Cystatin C is a protein from the family of cysteine proteinase inhibitors and is of interest as an early marker of decreased renal function. It is a protein that is synthesized at a constant rate by all cells containing nuclei, secreted into biological fluids: plasma, pleural, ascitic, cerebrospinal fluid, freely filtered through the glomerular membrane (due to its low molecular weight), fully metabolized in the kidneys, not secreted by the proximal renal tubules.

Renal resistive index (RRI) is a noninvasive instrument to evaluate kidney hemodynamics, and it is obtained by analysis of intrarenal arterial waves using Doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe pre-eclampsia and eclampsia.
* Polytraumatized patients.
* Patients admitted to ICU with sepsis.
* Both genders.
* Patients above 18 years.

Exclusion Criteria:

* patients known to have CKD.
* patients with congenital renal anomalies.
* patients with renal transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are admitted to SICU, Aswan university hospital, after polytrauma, pre-eclampsia, eclampsia and sepsis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Early detection of acute kidney injury. | Day 0,1,2,3,7
  Renal artery resistive index will be measured daily.Cystatin C will be measured on admission, after 24 hours and 72 hours.
Diagnosis of acute kidney injury. | Day 0,1,2,3,7
  Renal artery resistive index will be measured daily.Cystatin C will be measured on admission, after 24 hours and 72 hours.

SECONDARY OUTCOMES:
To grade the severity of AKI. | day 0,1,2,3,7
  Using the KDIGO criteria, AKI is staged as follows:
  Stage 1: Increase in serum creatinine to 1.5 to 1.9 times baseline, or increase in serum creatinine by ≥0.3 mg/dL, or reduction in urine output to <0.5 mL/kg/h for 6 to 12 h.
  Stage 2: Increase in serum creatinine to 2.0 to 2.9 times baseline, or reduction in urine output to <0.5 mL/kg/h for ≥12 h.
  Stage 3: Increase in serum creatinine to 3.0 times baseline, or increase in serum creatinine to ≥4.0 mg/dL, or reduction in urine output to <0.3 mL/kg/h for ≥24 h, or anuria for ≥12 h, or the initiation of renal replacement therapy, or, in patients <18 years, decrease in estimated glomerular filtration rate (eGFR) to <35 mL/min/1.73 m2.
To predict clinical outcome (clinical improvement) | Day 0,1,2,3,7,30
  To predict clinical outcome (clinical improvement) at 30 days
To predict clinical outcome (necessity for renal replacement therapy) | Day 0,1,2,3,7,30
  To predict clinical outcome (necessity for renal replacement therapy) at 30 days
To predict clinical outcome (death) | Day 0,1,2,3,7,30
  To predict clinical outcome (death) at 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Abolwafa, MSc, Principal Investigator — Aswan University; Ahmed E Abd Elrahman, MD, Principal Investigator — Sohag University
Locations (1):
- Aswan University, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pan HC, Yang SY, Chiou TT, Shiao CC, Wu CH, Huang CT, Wang TJ, Chen JY, Liao HW, Chen SY, Huang TM, Yang YF, Lin HY, Chan MJ, Sun CY, Chen YT, Chen YC, Wu VC. Comparative accuracy of biomarkers for the prediction of hospital-acquired acute kidney injury: a systematic review and meta-analysis. Crit Care. 2022 Nov 12;26(1):349. doi: 10.1186/s13054-022-04223-6. PMID 36371256
- [Background] Cruz EG, Broca Garcia BE, Sandoval DM, Gopar-Nieto R, Gonzalez Ruiz FJ, Gallardo LD, Ronco C, Madero M, Vasquez Jimenez E. Renal Resistive Index as a Predictor of Acute Kidney Injury and Mortality in COVID-19 Critically Ill Patients. Blood Purif. 2022;51(4):309-316. doi: 10.1159/000517469. Epub 2021 Jul 19. PMID 34280921
- [Background] Provenzano M, Rivoli L, Garofalo C, Faga T, Pelagi E, Perticone M, Serra R, Michael A, Comi N, Andreucci M. Renal resistive index in chronic kidney disease patients: Possible determinants and risk profile. PLoS One. 2020 Apr 1;15(4):e0230020. doi: 10.1371/journal.pone.0230020. eCollection 2020. PMID 32236125
- [Background] Fernando S, Polkinghorne KR. Cystatin C: not just a marker of kidney function. J Bras Nefrol. 2020 Mar;42(1):6-7. doi: 10.1590/2175-8239-JBN-2019-0240. Epub 2020 Apr 3. No abstract available. PMID 32255469